CLINICAL TRIAL: NCT00470028
Title: A Study of Transcranial Magnetic Stimulation (TMS) Treatment in Depressed Adolescents
Brief Title: Transcranial Magnetic Stimulation: Treatment Trial for Depressed Adolescents
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low recruitment.
Sponsor: The University of New South Wales (Other)
Collaborators: University of Sydney (Other); Monash University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04263
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-11

CONDITIONS: Depression
Keywords: TMS; Treatment; Adolescents; Safety; Efficacy
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation

SUMMARY:
This is a study to assess the effectiveness and safety of repetitive transcranial magnetic stimulation (rTMS) as a treatment for depressed 13-18 year olds.

In rTMS high-intensity, fluctuating magnetic fields non-invasively stimulate the cortex of the brain depolarizing neurons. No anesthetic is required and the treatment in subconvulsive. Recent studies suggest that rTMS can be an effective treatment for depressive illness in adults (Loo and Mitchell, 2005) and appears to be quite safe.

Minimal data of TMS use in adolescents psychiatric disorders. Data only existed in seven patients of the four that were depressed two showed improvement in their depression (Quintana, 2005). No sham-controlled studies have been conducted.

The investigators wish to assess this in a sham-controlled study of 30 adolescents. The investigators hypothesize that rTMS will have an antidepressant effect and produce no neuropsychological impairment.

DETAILED DESCRIPTION:
The study has two phases: the sham-controlled phase and an open phase.

Sham-controlled Phase

Participants are randomly assigned to an active or sham TMS condition.

Open Phase

Following the sham controlled period participants participants in the sham rTMS condition will be offered active rTMS. Participants will have the opportunity to receive up to 6 weeks of active rTMS.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Major Depressive Episode of no more then 3 years.
* Montgomery-Asberg Depression Rating Scale score of 20 or more.
* Aged between 13 and 18.
* May or may not be taking antidepressant medication.

Exclusion Criteria:

* Patient (or family is patient is under 18)not able to give informed consent.
* Failure to respond to ECT in current or past episodes of depression.
* Significant other Axis 1 psychiatric disorders e.g. schizophrenia.
* In imminent physical or psychological danger and needs a rapid clinical response due to inanition, psychosis or high suicide risk.
* Drug or alcohol abuse currently or in the last month.
* History of neurological illness e.g. epilepsy; neurosurgical procedure
* Mental in the cranium, a pacemaker, cochlear implant, medication pump or other electronic device.
* Women of child-bearing age whom pregnancy cannot be ruled out.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
All measures at baseline and at the end of each week of treatment in the blind phase and after every 2 weeks of treatment in the open phase.
Montgomery-Asberg Depression Rating Scale (MADRS)
Clinical Global Impressions Scale (CGI)

SECONDARY OUTCOMES:
All measures at baseline, at the end of the 4 week blind phase and at end of treatment in the open phase.
Rey Auditory Verbal Learning Test (RAVLT)
Digit span forwards and backwards and Digit symbols (WAIS)
Tower of London
Verbal Fluency
Trail A, B
Beck Depression Inventory
Centre for Epidemiological Studies - Depression - Child (CES-DC) scale

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, FRANZCP; MD, Principal Investigator — University of New South Wales
Locations (3):
- Australia (3):
  - Northside Clinic, Greenwich, New South Wales
  - Black Institute Building, School of Psychiatry, University of New South Wales, Sydney, New South Wales
  - Alfred Psychiatry Research Centre, The Alfred and Monash University Department of Psychological Medicine, The Alfred Hospital, Melbourne, Victoria

REFERENCES:
- [Result] Loo C, McFarquhar T, Walter G. Transcranial magnetic stimulation in adolescent depression. Australas Psychiatry. 2006 Mar;14(1):81-5. doi: 10.1080/j.1440-1665.2006.02251.x. PMID 16630205